CLINICAL TRIAL: NCT00688155
Title: Seniors Health and Activity Research Program-Pilot
Acronym: SHARP-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IA0133; 1R01AG029285-01 (NIH)
Record Dates: First submitted 2008-05-29; First posted 2008-06-02 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Cognitive Function
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned, with equal probability to one of four conditions: an educational control condition, moderate-intensity physical activity training, repetition lag cognitive training, or both physical activity and repetitive lag training.
Who Masked: Outcomes Assessor
Masking Description: Data collection related to study outcomes was performed by staff who were masked to intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical Activity Training (Experimental): The Physical Activity Training ((PAT) intervention consisted of center-based and home-based sessions comprised of aerobic, strength, flexibility, and balance training with a targeted duration of 150 mins/wk.
  Interventions: Behavioral: Physical Activity Training
- Cognitive Training (Experimental): The Cognitive Training (CT) intervention was developed to improve consciously-controlled memory processing or recollection of episodic memory information.
  Interventions: Behavioral: Cognitive Training
- Combined Intervention (Experimental): The Combined Intervention (PACT) was designed so that participants received both cognitive and physical activity training on the same day.
  .
  Interventions: Behavioral: Physical Activity Training; Behavioral: Cognitive Training
- Healthy Aging Education (Active Comparator): The Healthy Aging Education control intervention consisted of weekly lectures based on health education.
  Interventions: Behavioral: Healthy Aging Education

INTERVENTIONS:
Behavioral: Physical Activity Training — Two 1-hour center and two 15- to 45-minute home-based training sessions per week to include aerobic, strength, flexibility, and balance training for 6 months. The ultimate goal is to accumulate 150 minutes of walking per week between center and home-based sessions.
  Arms: Combined Intervention; Physical Activity Training
Behavioral: Cognitive Training — Two 1-hour sessions per week for the first two months and then one 1-hour session per week for months 3-6.
  Arms: Cognitive Training; Combined Intervention
Behavioral: Healthy Aging Education — One 1-hour lecture each week for 3 months, then monthly.
  Other Names: Healthy Aging
  Arms: Healthy Aging Education

SUMMARY:
The purpose of this pilot study is to develop and conduct well-designed trial to assess whether a multi-factorial intervention involving physical activity and cognitive training reduces the risk of significant cognitive decline in older individuals.

DETAILED DESCRIPTION:
Evidence from small or uncontrolled studies indicates that physical exercise and cognitive training have considerable promise as prevention strategies, to the extent that they are often recommended; however, their efficacy has not been established by an adequately powered randomized clinical trial.

This pilot study will provide the experience and data to assess whether physical activity and cognitive training separately improve cognitive function over 6 months. It will also determine whether a combination intervention holds promise beyond individual interventions without compromising adherence, and will provide information necessary to design a well-organized and efficient full scale, multi-center randomized clinical trial.

The Physical Activity Training (PAT) will consist of center-based and home-based sessions to include aerobic, strength, flexibility, and balance training. The actual time spent exercising will vary from person to person and will also vary depending on what stage of the study they are in.

The Cognitive Training (CT) intervention was developed to improve consciously-controlled memory processing or recollection of episodic memory information and produces changes in performance that transfer to executive function, such as working memory, planning and memory monitoring, as well as long term item memory and cognitive processing speed.

The Healthy Aging Education (HAE) control will combine health education-based lectures with light stretching and toning. HAE will include an experiential component, in which participants will learn how to take charge of their health and seek out appropriate medical services and information. Topics such as medications, foot care, traveling and nutrition will be covered.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 to 85 years
* Summary score between 88 (80 for less than 8 years of education) and 95 on the Modified Mini-Mental Exam
* Sedentary lifestyle, i.e., not actively participating in a formal exercise program within the past 3 months (defined as 30 minutes or more of formal exercise at least once a week; brisk walks will be considered formal exercise, leisurely walks will not)
* Fluency in standard American English (to limit staffing and translation costs in this pilot)
* Willingness to be randomized to any of the four intervention conditions

Exclusion Criteria:

* Failure to provide the name of a personal physician
* Living in a nursing home; persons living in assisted or independent housing will not be excluded
* Unable to communicate because of severe hearing loss or speech disorder
* Severe visual impairment, which would preclude completion of the assessments and/or intervention
* Neurologic disease, e.g. Alzheimer's (or other types of dementia), stroke that required hospitalization, Parkinson's, multiple sclerosis, amyotrophic lateral sclerosis, or prior diagnosis of mild cognitive impairment (MCI)
* Abnormal functioning based on the modified Telephone Interview for Cognitive Status (less than 30)
* Positive screen for MCI or dementia
* Scores greater than or equal to 1.5 standard deviations below normal on memory and non-memory domain tests (speed of processing, and verbal fluency)
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, active inflammatory disease
* Terminal illness with life expectancy less than 8 months, as determined by a physician
* Severe pulmonary disease, e.g., on home oxygen or chronic steroids
* Severe cardiac disease, including New York Health Association Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest which required resuscitation, use of a cardiac defibrillator, or uncontrolled angina
* Other significant co-morbid disease that would impair ability to participate in the exercise-based intervention, e.g. renal failure on hemodialysis, severe or acute psychiatric disorder (e.g. bipolar disorder or major depression, schizophrenia), excessive alcohol use (more than 14 drinks per wk); persons with managed depression (on stable dosage for at least 3 months) will not be excluded
* Baseline Geriatric Depression Scale score greater than 6
* Other significant factors that may affect the ability for cognitive training, including a history of head trauma resulting in a loss of consciousness, current use of benzodiazepines, hypnotic or anticholinergic agents, and current use of cognitive enhancing prescription or investigational medications (e.g., donepezil, selegiline, tacrine)
* Member of household is already enrolled
* Lives distant from the study site or is planning to move out of the area in next 3 years or leave the area for more than 3 months during the next year
* History of participation in a cognitive program in the last 2 years (includes research studies involving memory training)
* Myocardial infarction, coronary artery bypass graft, or valve replacement within past 6 months
* Serious conduction disorder (e.g., 3rd degree heart block), uncontrolled arrhythmia
* Pulmonary embolism or deep venous thrombosis within past 6 months
* Stroke, hip fracture, hip or knee replacement, or spinal surgery within past 4 months
* Receiving physical therapy for gait, balance, or other lower extremity training
* Severe hypertension, e.g., systolic blood pressure over 160 mmHg, diastolic blood pressure over 110 mmHg
* Other temporary intervening events, such as sick spouse, bereavement, or recent move
* Participation in another intervention trial; participation in an observational study may be permitted
* Inability to commit to intervention schedule requirements

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2009-06-30 (Actual); Study Completion 2010-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Espeland, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Available on request and development of a data sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: On request
Access Criteria: Data sharing agreement.

REFERENCES:
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Espeland MA, Rapp SR, Robertson J, Granek I, Murphy C, Albert M, Bassford T; Women's Health Initiative Memory Study. Benchmarks for designing two-stage studies using modified mini-mental state examinations: experience from the Women's Health Initiative Memory Study. Clin Trials. 2006;3(2):99-106. doi: 10.1191/1740774506cn140oa. PMID 16773952
- [Background] Legault C, Jennings JM, Katula JA, Dagenbach D, Gaussoin SA, Sink KM, Rapp SR, Rejeski WJ, Shumaker SA, Espeland MA; SHARP-P Study Group. Designing clinical trials for assessing the effects of cognitive training and physical activity interventions on cognitive outcomes: the Seniors Health and Activity Research Program Pilot (SHARP-P) study, a randomized controlled trial. BMC Geriatr. 2011 May 26;11:27. doi: 10.1186/1471-2318-11-27. PMID 21615936
- [Background] Espeland MA, Katula JA, Rushing J, Kramer AF, Jennings JM, Sink KM, Nadkarni NK, Reid KF, Castro CM, Church T, Kerwin DR, Williamson JD, Marottoli RA, Rushing S, Marsiske M, Rapp SR; LIFE Study Group. Performance of a computer-based assessment of cognitive function measures in two cohorts of seniors. Int J Geriatr Psychiatry. 2013 Dec;28(12):1239-50. doi: 10.1002/gps.3949. Epub 2013 Apr 16. PMID 23589390
- [Derived] Espeland MA, Rapp SR, Katula JA, Andrews LA, Felton D, Gaussoin SA, Dagenbach D, Legault C, Jennings JM, Sink KM; SHARP-P Study Group. Telephone interview for cognitive status (TICS) screening for clinical trials of physical activity and cognitive training: the seniors health and activity research program pilot (SHARP-P) study. Int J Geriatr Psychiatry. 2011 Feb;26(2):135-43. doi: 10.1002/gps.2503. PMID 21229597

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity Training: The Physical Activity Training ((PAT) intervention consisted of center-based and home-based sessions comprised of aerobic, strength, flexibility, and balance training with a targeted duration of 150 minutes/week. It included two center and two home-based training sessions per week for four months. Its primary focus was walking with the explicit intent of improving cardiovascular fitness. Other forms of endurance activity (e.g., stationary cycling) were used when regular walking was contraindicated for medical or behavioral reasons. Center-based physical activity sessions were supplemented with additional tailored home-based walking sessions at 1-2 per week during the first month.
  Physical Activity Training (PAT): Two 1-hour center and two 15- to 45-minute home-based training sessions per week to include aerobic, strength, flexibility, and balance training for 6 months. The ultimate goal is to accumulate 150 minutes of walking per week between center and home-based sessions.
- Cognitive Training: The Cognitive Training (CT) intervention was developed to improve consciously-controlled memory processing or recollection of episodic memory information. Sessions were center-based, conducted via computer, carried out with small groups, and monitored by skilled trainers. Training consisted of four consecutive 10-12 min sessions per day, administered two times per week for two months, which then tapered to one time per week for two additional months. For each session, participants studied a list of 30 words, followed by a recognition test consisting of the 30 studied words and 30 new words with each new word repeated once, and asked to respond "yes" to study words and "no" to the new items both times they occurred.
  Cognitive Training (CT): Two 1-hour sessions per week for the first two months and then one 1-hour session per week for months 3-6.
- Combined Intervention: The Combined Intervention (PACT) was designed so that participants received both cognitive and physical activity training on the same day. To avoid the potential impact of physical fatigue on cognitive training, the cognitive treatment was delivered prior to the physical activity treatment. It included both the PA and CT interventions.
  Physical Activity Training (PAT): Two 1-hour center and two 15- to 45-minute home-based training sessions per week to include aerobic, strength, flexibility, and balance training for 6 months. The ultimate goal is to accumulate 150 minutes of walking per week between center and home-based sessions.
  Cognitive Training (CT): Two 1-hour sessions per week for the first two months and then one 1-hour session per week for months 3-6.
- Healthy Aging: The Healthy Aging Education control intervention consisted of weekly lectures based on health education and was based on a program developed by the Lifestyle Interventions and Independence for Elders pilot trial [Rejeski, 2005; Lifestyle Interventions and Independence for Elders, 2006]. Topics such as medications, foot care, traveling and nutrition were covered. The purpose of the intervention was to provide contact time with participants.
  Healthy Aging Education (HAE): One 1-hour lecture each week for 3 months, then monthly.
Period: Overall Study
Arm/Group | Physical Activity Training | Cognitive Training | Combined Intervention | Healthy Aging
Started | 18 | 18 | 19 | 18
Completed | 16 | 16 | 18 | 17
Not Completed | 2 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Aging: The Healthy Aging Education control intervention consisted of weekly lectures based on health education and was based on a program developed by the Lifestyle Interventions and Independence for Elders pilot trial [Rejeski, 2005; LIFE, 2006]. Topics such as medications, foot care, traveling and nutrition were covered. The purpose of the intervention was to provide contact time with participants.
  Healthy Aging Education (HAE): One 1-hour lecture each week for 3 months, then monthly.
- Total: Total of all reporting groups
Arm/Group | Physical Activity Training | Cognitive Training | Combined Intervention | Healthy Aging | Total
Number analyzed (Participants) | 18 | 18 | 19 | 18 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.5 (4.8) | 76.0 (5.2) | 76.9 (4.0) | 75.4 (4.8) | 76.4 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 12 | 7 | 37
  Male | 8 | 10 | 7 | 11 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 1 | 1 | 4 | 1 | 7
  Caucasian | 17 | 17 | 15 | 17 | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 19 | 18 | 73
400 meter walk time [Mean (Standard Deviation); unit: Seconds] | 360 (48) | 331 (50) | 347 (56) | 331 (66) | 342 (55)
Modified MiniMental State Exam Score [Mean (Standard Deviation); unit: Units on a scale] — The Modified Mini Mental State Exam (3MS) Memory Functioning questionnaire asks the participant to rate on a scale of 1 (always) to 7 (never) how often remembering something presents a problem. In order to participate, subjects had to score at least an 88 or greater if their education level is greater than 8 years and if education level was 0-8 years, scores had to be at least an 80 or higher. The possible scores (units on a scale) range from 0 to 100, with higher scores reflecting better global cognitive functioning.
  Units on a scale | 94.6 (3.9) | 95.6 (3.4) | 94.6 (4.3) | 94.3 (2.4) | 94.8 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Composite Cognitive Function in Z-scores (i.e. Which Converts Raw Data to Standard Deviation (SD) Units: [Score-mean]/SD]). This Composite is Formed by Averaging the Z-scores From Individual Tests.
Description: 6 measures of executive functioning: Self-Ordered Pointing task (24): working memory
  1- and 2-Back tests (25-26): working memory Eriksen flanker (27): response inhibition Task Switching (28): attentional flexibility Trail Making (29): executive function z-score=(raw score-mean)/standard deviation 4 measures of episodic memory Hopkins Verbal Learning Test (30) Wechsler Memory Scale-III (31)
  A composite of 10 scores: dividing each's difference from the baseline mean by the baseline SD, averaging the 6 executive function and 4 episodic memory z-transformed measures, and norming to have SD 1.
  24. Petrides. Neuropsych 1982;20:249-62. 25. Dobbs. Psychol Aging 1989;4:500-3. 26. Jonides. J Cog Neurosci 1997;9:462-75. 27. Ericksen. Br J Sports Med 2009;43:22-4. 28. Kramer. Acta Psychologica 1999;101:339-78. 29. Reitan. Per Motor Skills 1958;8:271-6. 30. Brandt. Clin Neuropsych 1991;5:125-42. 31. Wechsler D.1997. Psychological Corporation, Harcourt, Inc: San Antonio.
Time Frame: Changes from baseline at 4 months in z-scores.
Population: Participants assessed at four months post-randomization. Note that this does not include all who were randomized due to dropout.
Measure: Mean (Standard Error); unit: z-scores (e.g.Standard Deviation Units)
Arm/Group | Physical Activity Training | Cognitive Training | Combined Intervention | Healthy Aging
Number analyzed (Participants) | 16 | 16 | 19 | 17
z-scores (e.g.Standard Deviation Units) | 0.71 (0.18) | 0.62 (0.18) | 0.71 (0.17) | 0.65 (0.18)
Statistical Analysis 1: Comparison: Healthy Aging; Marginal comparisons of physical activity training vs no physical activity training; Test type: Equivalence — Two-sided test of mean differences from baseline; p = 0.66, ANOVA — Physical activity training versus no physical activity training;; Mean Difference (Net) = 0.08, Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Healthy Aging; Marginal comparisons of physical activity training versus no physical activity training; Test type: Equivalence — Two-sided tests of mean differences from baseline; p = 0.55, ANOVA — P-value for physical activity training is 0.55; Mean Difference (Final Values) = -0.06, Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Cognitive Training; Marginal comparisons of cognitive training versus no cognitive training; Test type: Equivalence — Two Sided Test of Mean Difference from baseline; p = 0.95, ANOVA; Mean Difference (Net) = 0.02, Standard Error of Mean 0.25
Statistical Analysis 4: Comparison: Cognitive Training; Marginal comparisons of cognitive training versus no cognitive training; Test type: Equivalence — Two Sided Test of Mean Difference from baseline; p = 0.48, ANOVA; Mean Difference (Net) = 0.07, Standard Error of Mean 0.26

2. Secondary Outcome: Change in Executive Function: Z-score Formed by Averaging the Individual Z-scores From the Five Tests Listed Below.
Description: Composite of 5 tasks:
  Self-Ordered Pointing Task of planning, working memory, and monitoring. Subjects view 16 abstract shapes and choose a shape so that each is selected by the 16th trial and none is chosen more than once. (Eriksen, Percept Psychophysiology 1974;16:143-49).
  N-Back Test of working memory. Subjects see individual letters and indicate whether the letter is the same as the nth back letter, with n equal to 1 and 2. (Dobbs, Psychol Aging 1989;4:500-3.)
  Eriksen flanker task of response incompatibility. Subjects see an arrow facing either right or left and indicate the direction.The target displays can be neutral congruent, or incongruent. (Eriksen, Percept Psychophys 1974;16:143-49.)
  Trail Making Test-Part B of alternating attention. Subjects connect 25 labeled circles and are scored by completion time. The lower the scores the better the performance. See details in the primary outcome.
  Raw scores for each test were converted to z-scores.
Time Frame: Baseline to 4 months
Population: Participants assessed at 4 months -- note some dropouts occurred
Measure: Mean (Standard Error); unit: z-scores (e.g. SD units)
Arm/Group | Physical Activity Training | Cognitive Training | Combined Intervention | Healthy Aging
Number analyzed (Participants) | 16 | 16 | 19 | 17
z-scores (e.g. SD units) | 0.32 (0.19) | 0.58 (0.19) | 0.60 (0.18) | 0.58 (0.19)

3. Secondary Outcome: Composite Episodic Memory
Description: Composite of 4 components.
  The Hopkins Verbal Learning Test (HVLT) of verbal learning. Subjects hear 12 words and repeat as many as possible. This is repeated twice for a total of 3 trials. 20 mins later the subject is asked to recall as many words as possible. Subjects also do a recognition trial with 24 words. Scores for immediate and delayed recall, and recognition are calculated.(Brandt J. Clin Neuropsych 1991;5:125-42).
  The Logical Memory (LM) test The LM test has 2 parts. In Part 1, subjects hear a story and recall as many pieces as possible immediately and after a 30 minute delay. Subjects receive a story unit score for accuracy of re-telling story details and a thematic score for recalling story themes. The higher the scores the better the performance. ( Wechsler D. The Wechsler Memory Scale-3rd Edition (WHM-III). Psycholog Corp, Harcourt, Inc.)
  Individual scores are converted to z-scores and averaged to form the composite.
Time Frame: Change a 4 months
Population: Participants assessed at 4 months
Measure: Mean (Standard Error); unit: z-scores (e.g. SD units)
Arm/Group | Physical Activity Training | Cognitive Training | Combined Intervention | Healthy Aging
Number analyzed (Participants) | 16 | 16 | 19 | 17
z-scores (e.g. SD units) | 0.84 (0.21) | 0.42 (0.21) | 0.56 (0.20) | 0.47 (0.21)
Statistical Analysis 1: Comparison: Healthy Aging; Marginal comparisons of physical activity training versus no physical activity training; Test type: Equivalence — Two-sided tests of marginal means; p = 0.23, ANOVA; Mean Difference (Final Values) = 0.26, Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Cognitive Training; Marginal comparisons of cognitive training versus no cognitive training; Test type: Equivalence — Two Sided Test of Mean Difference from baseline; p = 0.42, ANOVA; Mean Difference (Net) = -0.16, Standard Error of Mean 0.29

ADVERSE EVENTS:
Time Frame: 4 months. Note that all randomized participants are included in the adverse events accounting. Only a subset are included in the analyses of outcomes - -these by protocol were limited to those providing outcome data.
Description: Clinicaltrials.gov definition was used.
  A Data Safety Monitoring Board (DSMB) monitored all aspects of the study, including those that require access to blinded data. Included in each DSMB report was a summary of any safety issues that may have arisen since the last DSMB meeting, prepared by the Safety Officer. Any serious adverse event that might be due to the study intervention was to be reported immediately to the DSMB, the Institutional Review Board (IRB) and the Project Office.
Arm/Group | Physical Activity Training | Cognitive Training | Combined Intervention | Healthy Aging
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/18 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 8/18 | 5/18 | 6/19 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity Training (N=18) | Cognitive Training (N=18) | Combined Intervention (N=19) | Healthy Aging (N=18)
Stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — The stoke occurred after randomization but prior to any intervention delivery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity Training (N=18) | Cognitive Training (N=18) | Combined Intervention (N=19) | Healthy Aging (N=18)
Non-serious (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (5) | 6 (6) | 1 (1) — There have been 22 Adverse Events reported, e.g. knee/hip/shin pain, back pain, nose bleeds, high blood pressure, shortness of breath, headaches, falls, diverticulitis, ankle and toe injuries, etc. Records no longer exist for greater specificity.

LIMITATIONS AND CAVEATS:
While large enough to meet its objectives, our pilot trial involved a modest sample size and short follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No